CLINICAL TRIAL: NCT05493280
Title: Quantifying Hyperpigmentation Response to Fractionated 1927nm in Fitzpatrick Skin Phototype V and VI: A Pilot Study
Brief Title: Fractionated 1927nm Laser for Hyperpigmentation in Fitzpatrick Skin Phototypes V and VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Principle Investigator, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0672
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Participants- Pre-Ttreatment Only (Other): Subjects who are interested in treatment for hyperpigmentation will be enrolled for this study.
  Subjects will be pre-treated with tretinoin/hydroquinone prior to treatments. No post-treatment care.
  Interventions: Device: MOXI
- Healthy Participants- Post-Treatment Only (Other): Subjects who are interested in treatment for hyperpigmentation will be enrolled for this study.
  Subjects will wash out of any topical medications and will receive treatment. Post-treatment care will include use of temovate for 4 days.
  Interventions: Device: MOXI

INTERVENTIONS:
Device: MOXI — Patients will receive treatment using f1927 devices and will be treated over the affected areas, once each month for a total of three months.

SUMMARY:
The primary objective of this study is to assess the efficacy of 1927nm non-ablative fractionated laser therapy to treat hyperpigmentation in patients ages 18-75 with Fitzpatrick Skin Phototypes V and VI and explore an effective, adjunctive pre- and post-procedural regimen to prevent iatrogenic dyspigmentation or scarring in this population.

DETAILED DESCRIPTION:
This single-center clinical trial is being conducted over the course of 7 months, including one Initial Screening Visit (-42 to -28 Days) and three treatments (Day 0, Day 30, Day 60) followed by 1-month and 3-month follow-up visits (Day 90 and Day 120). The primary objective of this study is to assess the efficacy of 1927nm non-ablative fractionated laser therapy to treat hyperpigmentation in patients ages 18-75 with Fitzpatrick Skin Phototypes V and VI and explore an effective, adjunctive pre- and post-procedural regimen to prevent iatrogenic dyspigmentation or scarring in this population.

The Investigators will explore this question with a non-blinded, pilot study at a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, female, and non-binary adults between 18 and 75 years of age
2. Fitzpatrick Skin Phototype V and VI
3. Individuals deemed by the Investigator to have clinically significant hyperpigmentation on their face and desire treatment and correction of this condition
4. Individuals willing to withhold aesthetic therapies (excluding those explicitly prescribed by the Investigator as pre-treatment) for the duration of the study
5. Women of childbearing potential who agree to take a urine pregnancy test at the Screening visit or when deemed by Investigator. Women of childbearing potential must have a negative urine pregnancy test and must not be lactating at Screening. Women must be willing and able to use an acceptable method of birth control (see below) during the study. Women will not be considered of childbearing potential if one or more of the following is documented:

   * Postmenopausal for 12 months prior to initiation of the study
   * Without a uterus +/- both ovaries prior to initiation of the study
   * Bilateral tubal ligation 6 months prior to initiation of the study
6. Individuals of childbearing potential who use an acceptable method of contraception for the duration of the study. Acceptable modes of birth control include the following:

   * Established use of hormonal contraception (oral, injectable, implanted, patch or vaginal ring)
   * Barrier methods with spermicide: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
   * Intrauterine device (IUD) or intrauterine system (IUS)
   * Surgical sterilization (e.g., vasectomy confirmed to be effective by sperm count check, tubal occlusion, hysterectomy, bilateral salpingectomy/oophorectomy)
   * Abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal methods are not acceptable forms of contraception.
7. Individuals who can read, speak, write, and understand English and who are willing to provide written informed consent.
8. Individuals willing to sign a photography release.
9. Individuals willing and able to cooperate with all study requirements for the duration of the study, including prescribed pre- and post-procedure topical regimens

Exclusion Criteria:

1. Ages < 18 or > 75 years old
2. Fitzpatrick Skin Phototypes I-IV
3. Known history of allergies or irritant contact dermatitis in response to general skin care products, including Hydroquinone and Retinol
4. Known allergies or irritant contact dermatitis in response to common ingredients of physical sunscreen, including but not limited to Zinc Oxide
5. Known allergies or irritant contact dermatitis to topical anesthetics, including Benzocaine and Tetracaine.
6. Active local or systemic disorders that may affect wound healing or integrity of the integumentary system
7. History of active or inactive systemic granulomatous disease, (e.g., Sarcoidosis, Tuberculosis, Granulomatosis with Polyangiitis, etc.), or connective tissue disorders (e.g., Systemic Lupus Erythematosus, Dermatomyositis, Scleroderma, etc.)
8. Recent history of surgery or significant trauma to the area(s) to be treated
9. Significant scarring (excluding acne scars) in the area(s) to be treated
10. Current or history of hypertrophic scarring or keloid scars
11. Severe or cystic and clinically active acne on the area(s) to be treated
12. Tattoos in the area(s) to be treated
13. Individuals who currently have cancerous or pre-cancerous lesions in the area(s) to be treated and/or have a history of skin cancer
14. Individuals with skin pathology and/or pre-existing dermatologic condition in the treatment area (i.e., psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation) that the Investigator deems inappropriate for participation or could interfere with outcomes of the study.
15. History of chronic drug or alcohol use.
16. Microdermabrasion or glycolic acid treatment to the treatment area(s) within 4 weeks of study participation or who plan on having this treatment during the study.
17. History of the following cosmetic treatments in the area(s) to be treated:

    * Injectable filler of any type within the past 2 weeks
    * Neurotoxins within the past week
    * Ablative resurfacing laser treatment within the past 6 months
    * Non-ablative, rejuvenating laser or light treatment within the past 6 months
    * Chemical peel or dermabrasion within the past 3 months
18. Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study devices:

    • Antiplatelet agents/anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use), and/or
19. Psychiatric drugs that, in the Investigator's opinion, would impair the subject from understanding protocol requirements or understanding and signing consent.
20. Individuals who are pregnant or nursing or those planning on becoming pregnant during the study according to self-report.
21. Immunocompromised individuals or those currently using immunosuppressive medications and/or radiation.
22. Individuals with uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension, or hypothyroidism. Those with multiple health conditions may still be excluded from participation even if conditions are controlled.
23. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures planned during the study.
24. Individuals who, in the Investigator's opinion, have a history of poor cooperation, unreliability or noncompliance with medical treatment.
25. Individuals who are unable to understand instructions or give informed consent
26. Individuals who have physical or psychological conditions which, in the opinion of the Investigator, makes them unable to complete the study per protocol (e.g., not likely to avoid other cosmetic treatments to area; not likely to stay in study for entire duration due to other commitments; or those with concomitant conditions that may develop symptoms that might confuse or confound study treatments or assessments).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — UT Southwestern- Department of Plastic Surgery
Locations (1):
- UT Southwestern Medical Center- Dept of Plastic Surgery, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 10 subjects who completed Part 1 (Pre-Treatment Group), only 6 continued to washout and Part 2 portion of this study and thus additional subjects were enrolled in part 2 (Post-Treatment Group) as represented in the data table below.
Groups:
- Healthy Subjects: First Pre-Treatment Only(Part 1), then Post-Treatment Only(Part 2) after washout: Part 1: Subjects will be pre-treated with tretinoin/hydroquinone prior to treatments. No post-treatment care.
  Subjects will wash out of any topical medications for at least 6 weeks.
  Part 2: Care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
- Healthy Participants: Post-Treatment- Part 2 Only: Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Period: Part 1 Intervention (7 months)
Arm/Group | Healthy Subjects: First Pre-Treatment Only(Part 1), then Post-Treatment Only(Part 2) after washout | Healthy Participants: Post-Treatment- Part 2 Only
Started | 12 | 0
Completed | 10 | 0
Not Completed | 2 | 0
Period: Washout Period (1 month)
Arm/Group | Healthy Subjects: First Pre-Treatment Only(Part 1), then Post-Treatment Only(Part 2) after washout | Healthy Participants: Post-Treatment- Part 2 Only
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0
Period: Part 2 intervention (7 months)
Arm/Group | Healthy Subjects: First Pre-Treatment Only(Part 1), then Post-Treatment Only(Part 2) after washout | Healthy Participants: Post-Treatment- Part 2 Only
Started | 6 (6 subjects from Part 1 continued to Part 2) | 3 (3 additional subjects who were not on part 1 were enrolled in Part 2)
Completed | 5 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 12 subjects started Part 1 (Pre-Treatment Group), and after washout, in Part 2 portion of this study, 3 additional subjects were enrolled as represented in the table below.
Groups:
- Healthy Subjects: First Pre-Treatment Only(Part 1), Then Post-Treatment Only(Part 2) After Washout: Part 1: Subjects will be pre-treated with tretinoin/hydroquinone prior to treatments. No post-treatment care.
  Part 2: Care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
- Healthy Participants: Part 2 Only: Subjects will wash out of any topical medications and will receive 3 treatments. Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive treatment using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects: First Pre-Treatment Only(Part 1), Then Post-Treatment Only(Part 2) After Washout | Healthy Participants: Part 2 Only | Total
Number analyzed (Participants) | 12 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 3 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 subject in Group 2 withdrew consent after Part 1 Intervention
  Participants
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 11 | 1 | 12
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 0 | 10
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Spots - Front of Face (Part 1)
Description: Quantitively assessment of change in overall spots using measurements provided VISIA 3D analysis of front face
  Count- the number of individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: spots
Groups:
- Healthy subjects-Part 1:- Pre-Treatment Only: Part 1: Subjects will be pre-treated with tretinoin/hydroquinone prior to treatments. No post-treatment care.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Arm/Group | Healthy subjects-Part 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
spots
  Baseline | 53.60 (14.01)
  1 Month | 58.47 (13.73)
  3 Months | 56.44 (15.14)

2. Primary Outcome: Change in Spots - Front of Face (Part 2)
Description: as for outcome 1
Time Frame: Baseline, 1 Month and 3 Months
Population: Data from 6 subjects in Part 1 who continued to Part 2 after washout and 2 new subjects who were added to Part 2 portion of this study were analyzed and reported in the data table below. 1 subject from Part 2, withdrew consent after 1st treatment and didn't return for 2nd treatment visit. So this subject's data wasn't included in the analysis.
Measure: Mean (Standard Deviation); unit: spots
Groups:
- Healthy subjects-Part 2- Post-Treatment Only: Part 2: Subjects will wash out of any topical medications and will receive 3 treatments. Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Arm/Group | Healthy subjects-Part 2- Post-Treatment Only
Number analyzed (Participants) | 8
spots
  Baseline | 56.57 (15.68)
  1 Month | 56.45 (18.40)
  3 Months | 49.93 (21.38)

3. Primary Outcome: Change in Spots- Left Side of Face (Part 1)
Description: Quantitively assessment of change in overall spots using measurements provided VISIA 3D analysis of left side of face
  Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: spots
Groups:
- Group 1:- Pre-Treatment Only: Part 1: Subjects will be pre-treated with tretinoin/hydroquinone prior to treatments. No post-treatment care.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
spots
  Baseline | 50.90 (13.22)
  1 Month | 49.37 (14.37)
  3 Months | 45.88 (11.26)

4. Primary Outcome: Change in Spots- Left Side of Face (Part 2)
Description: as for outcome 3
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: spots
Groups:
- Healthy subjects- Part 2- Post-Treatment Only: Part 2: Subjects will wash out of any topical medications and will receive 3 treatments. Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Arm/Group | Healthy subjects- Part 2- Post-Treatment Only
Number analyzed (Participants) | 8
spots
  Baseline | 48.01 (17.18)
  1 Month | 43.78 (13.07)
  3 Months | 41.94 (17.03)

5. Primary Outcome: Change in Spots- Right Side of Face (Part 1)
Description: Quantitively assessment of change in overall spots using measurements provided VISIA 3D analysis of right side of face
  Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
spots
  Baseline | 46.49 (14.05)
  1 Month | 46.47 (15.27)
  3 Months | 46.15 (13.68)

6. Primary Outcome: Change in Spots- Right Side of Face (Part 2)
Description: as for outcome 5
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: spots
Groups:
- Group 2- Post-Treatment Only: Part 2: Subjects will wash out of any topical medications and will receive 3 treatments. Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
spots
  Baseline | 41.65 (15.69)
  1 Month | 44.87 (16.62)
  3 Months | 43.68 (13.83)

7. Primary Outcome: Change in UV Spots- Front of Face (Part 1)
Description: Quantitively assessment of change in overall UV spots using measurements provided VISIA 3D analysis of front side of face Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: UV Spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
UV Spots
  Baseline | 4.55 (6.36)
  1 Month | 4.26 (5.94)
  3 Months | 3.67 (6.92)

8. Primary Outcome: Change in UV Spots- Front of Face (Part 2)
Description: as for outcome 7
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: UV Spots
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
UV Spots
  Baseline | 6.01 (6.28)
  1 Month | 7.92 (9.86)
  3 Months | 4.70 (5.91)

9. Primary Outcome: Change in UV Spots- Left of Face (Part 1)
Description: Quantitively assessment of change in overall UV spots using measurements provided VISIA 3D analysis of left side of the face
  Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: UV Spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
UV Spots
  Baseline | 5.87 (5.90)
  1 Month | 4.69 (5.17)
  3 Months | 5.69 (10.54)

10. Primary Outcome: Change in UV Spots- Left of Face (Part 2)
Description: as for outcome 9
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: UV Spots
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
UV Spots
  Baseline | 4.60 (8.01)
  1 Month | 2.50 (3.71)
  3 Months | 3.54 (3.30)

11. Primary Outcome: Change in UV Spots- Right Side if Face (Part 1)
Description: Quantitively assessment of change in overall UV spots using measurements provided VISIA 3D analysis of right side of face
  Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: UV Spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
UV Spots
  Baseline | 6.35 (7.58)
  1 Month | 4.25 (4.34)
  3 Months | 4.51 (6.32)

12. Primary Outcome: Change in UV Spots- Right Side if Face (Part 2)
Description: as for outcome 11
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: UV Spots
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
UV Spots
  Baseline | 2.71 (3.43)
  1 Month | 3.33 (3.32)
  3 Months | 3.50 (3.27)

13. Primary Outcome: Change in Brown Spots- Front of Face (Part 1)
Description: Quantitively assessment of change in overall UV spots using measurements provided VISIA 3D analysis of front of face
  Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: Brown Spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
Brown Spots
  Baseline | 35.14 (10.73)
  1 Month | 34.31 (12.29)
  3 Months | 32.73 (20.67)

14. Primary Outcome: Change in Brown Spots- Front of Face (Part 2)
Description: as for outcome 13
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Brown Spots
Groups:
- Group 2- Post-Treatment Only: Subjects will wash out of any topical medications and will receive 3 treatments. Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive treatment using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
Brown Spots
  Baseline | 27.67 (6.31)
  1 Month | 39.74 (14.29)
  3 Months | 33.36 (14.79)

15. Primary Outcome: Change in Brown Spots- Left of Face (Part 1)
Description: Quantitively assessment of change in overall UV spots using measurements provided VISIA 3D analysis of left side of face
  Count= the number if individual features detected in the region of interest.
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: Brown spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
Brown spots
  Baseline | 47.87 (14.20)
  1 Month | 47.97 (20.96)
  3 Months | 45.81 (13.97)

16. Primary Outcome: Change in Brown Spots- Left of Face (Part 2)
Description: as for outcome 15
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Brown spots
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
Brown spots
  Baseline | 39.03 (18.95)
  1 Month | 45.10 (14.16)
  3 Months | 39.49 (14.55)

17. Primary Outcome: Change in Brown Spots- Right Side of Face (Part 1)
Description: as for outcome 11
Time Frame: Baseline, 1 Month and 3 Months
Population: Subjects who completed Part 1 intervention are only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: Brown Spots
Arm/Group | Group 1:- Pre-Treatment Only
Number analyzed (Participants) | 10
Brown Spots
  Baseline | 41.73 (15.87)
  1 Month | 47.59 (13.77)
  3 Months | 41.42 (15.08)

18. Primary Outcome: Change in Brown Spots- Right Side of Face (Part 2)
Description: as for outcome 11
Time Frame: Baseline, 1 Month and 3 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Brown Spots
Arm/Group | Group 2- Post-Treatment Only
Number analyzed (Participants) | 8
Brown Spots
  Baseline | 33.83 (11.95)
  1 Month | 34.27 (19.96)
  3 Months | 40.99 (7.26)

ADVERSE EVENTS:
Time Frame: 3 Months
Description: For 1 subject in Part 2, AEs were collected until they withdrew consent [i.e., after 1st treatment (2nd visit)]
Groups:
- Part 1 Intervention: Part 1: Subjects will be pre-treated with tretinoin/hydroquinone prior to treatments. No post-treatment care.
  Part 2: Care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
- Part 2 Intervention (after Part 1): Subjects will wash out of any topical medications and will receive 3 treatments.
  Subjects will wash out of any topical medications and will receive 3 treatments. Post-treatment care will include use of temovate/ice for 4 days.
  MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
- Part 2 Intervention only: MOXI: Patients will receive 3 treatments using f1927 devices and will be treated over the affected areas, once each month for a total of three months.
  F1927 nm treatment and energy parameters included a pulse energy of 10 mJ, density of 10% with 10% coverage, and six total passes.
Arm/Group | Part 1 Intervention | Part 2 Intervention (after Part 1) | Part 2 Intervention only
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT05493280/Prot_SAP_000.pdf